CLINICAL TRIAL: NCT01495338
Title: A Comparison of the Safety and Comfort of AC-170
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aciex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-100-0013
Record Dates: First submitted 2011-12-15; First posted 2011-12-20 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Normal Ocular Health
MeSH Terms: interventions — Cetirizine; Olopatadine Hydrochloride; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AC-170 0.17% (Experimental)
  Interventions: Drug: AC-170 0.17%
- AC-170 0.24% (Formulation 1) (Experimental)
  Interventions: Drug: AC-170 0.24% (Formulation 1)
- AC-170 0.24% (Formulation 2) (Experimental)
  Interventions: Drug: AC-170 0.24% (Formulation 2)
- Olopatadine hydrochloride 0.2%/Tears Naturale II (Placebo Comparator)
  Interventions: Drug: Olopatadine hydrochloride 0.2%/Tears Naturale II

INTERVENTIONS:
Drug: AC-170 0.17% — 1 drop in one eye at one timepoint
  Arms: AC-170 0.17%
Drug: AC-170 0.24% (Formulation 1) — 1 drop in one eye at one timepoint
  Arms: AC-170 0.24% (Formulation 1)
Drug: AC-170 0.24% (Formulation 2) — 1 drop in one eye at one timepoint
  Arms: AC-170 0.24% (Formulation 2)
Drug: Olopatadine hydrochloride 0.2%/Tears Naturale II — 1 drop in one eye at one timepoint
  Arms: Olopatadine hydrochloride 0.2%/Tears Naturale II

SUMMARY:
The purpose of this study is to evaluate the safety and comfort of AC-170 compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to avoid the use of ocular medications or topical ocular preparations within protocol specific time period.

Exclusion Criteria:

* Known contraindications or sensitivities to the study medication or its components.
* Any ocular condition that, in the opinion of the investigator, could affect the subjects safety or trial parameters.
* Use of disallowed medications during the period indicated prior to the study enrollment or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Drop Comfort Score | during 3 minute period
  drop comfort on 0-10 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States